CLINICAL TRIAL: NCT02266225
Title: Measuring the Implementation of a Group-based Lifestyle-integrated Functional Exercise (Mi-LiFE) Intervention Delivered in Primary Care for Older Adults Aged 75 Years or Older: A Pilot Feasibility Study
Brief Title: Measuring the Implementation of the LiFE Program in Primary Care for Older Adults Aged 75 Years or Older
Acronym: Mi-LIFE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Waterloo (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Lora Giangregorio, Associate Professor, University of Waterloo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19377
Record Dates: First submitted 2014-09-10; First posted 2014-10-16 (Estimated); Results first posted 2019-08-19 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Chronic Disease
Keywords: Chronic disease management; Physical activity; Fall prevention; Strength and balance exercise
MeSH Terms: conditions — Chronic Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle-integrated functional exercise (Experimental): Lifestyle-integrated functional exercise- one individual and four group-based sessions led by a physiotherapist over two months, and two phone calls one week and one month following final group-based exercise session.
  Interventions: Other: Lifestyle-integrated Functional Exercise

INTERVENTIONS:
Other: Lifestyle-integrated Functional Exercise — Lifestyle-integrated functional exercise- one individual and four group-based sessions led by a physiotherapist over two months, and two phone calls one week and one month following final group-based exercise session.

SUMMARY:
The goal of this study is to evaluate how to implement an evidence-based lifestyle-integrated strength and balance exercise (LiFE) intervention in primary care to promote increased physical activity (PA) and improvements in function and quality of life in older adults 75 years or older. This study will evaluate the public health impact of the LiFE intervention using the RE-AIM model: reach (recruitment), effectiveness (PA levels), adoption (physician acceptance), implementation (fidelity), and maintenance (retention, adherence). If the intervention appears feasible, we will use the resultant information to design a larger pragmatic trial.

DETAILED DESCRIPTION:
Physical activity has numerous health and functional benefits for older adults, including increased lifespan, performing daily activities better, and improving quality of life. However, engaging older adults with multiple chronic diseases in traditional exercise programs is challenging. Community exercise programs may not meet the needs of frail older adults or be accessible because of physical limitations or travel required. Although structured, supervised exercise can be effective, it may not be realistic to implement on a population-wide basis. Although there is substantial evidence demonstrating that exercise can improve multiple health outcomes, there is limited research defining how exercise should be implemented in practice to engage older adults with chronic diseases.

Declines in person-centered outcomes (e.g., function, quality of life) and an increased risk of falls, cardiovascular events, and fractures occur with aging and may be amenable to interventions. Primary care is an ideal setting for identifying elderly patients in need of exercise intervention. However, a cost-effective, generalizable model of chronic disease management for older adults using exercise in this setting remains elusive. Further, the delivery of individualized exercise prescription for all older adults may not be feasible.

A recent study demonstrated that teaching older adults to integrate exercise into daily life activities was effective for reducing falls and improving function in older adult fallers. In addition, there is evidence that integrating balance and strength exercises into activities of daily living may promote long-term exercise participation, by "instituting new habitual behaviors within selected situational contexts that serve as prompts for action" . Therefore, the proposed physiotherapist-led group-based lifestyle-integrated functional exercise intervention delivered in primary care is timely. Recently announced changes to funding will allow physiotherapists to work within family health teams. However, there are no guidelines for how physiotherapy resources should be allocated.

This pilot feasibility study will evaluate how we can use these resources efficiently for chronic disease management in older adults via a novel intervention that teaches them lifestyle-integrated therapeutic exercise. The long-term aim is to improve the capacity for care providers in an interdisciplinary setting to offer patient-centered care that includes exercise to older adults 75 years or older. Thus, we propose to evaluate the pragmatic implementation of a group-based intervention in primary care that teaches older adults to integrate functional balance and strength exercises into daily activities as a relevant strategy, also known as the Lifestyle-integrated Functional Exercise (LiFE) program. The LiFE program is proposed as a strategy to engage older adults in sustainable exercise participation to improve chronic disease management and quality of life.

Our research objectives are related to feasibility, retention, and adherence and include: (1) to evaluate the number of participants we can recruit over 6 months: The intervention will be considered feasible if we recruit 32 participants over 6 months. Data collected from a screening program at the Centre for Family Medicine over 6 months shows that we have recruited 198 individuals who were not regularly exercising and 59 of those individuals agreed to receive information about exercise. Recruitment of 32 participants at one site over 6 months translates to 576 participants with 3 sites in three years; (2) to determine intervention retention rates: The intervention will be considered feasible if 75% of the sample complete the 6 month follow-up assessments; 3) to determine adherence to the exercise intervention: The intervention will be considered feasible if 50% of the participants complete balance and strength activities ≥3 days per week over the 6 month study period. Our criteria are based on randomized controlled trial data in exercise and falls prevention research showing that the completion of balance and strength exercise ≥ 3 times per week was positively associated with fall outcomes. In another study, the mean number of days in which the balance and strength activities were completed per week in the final month of the LiFE program was 3.89 of a maximum 7 days. Notably, a 47% adherence to the LiFE program over the first 6 months was associated with clinically relevant reduction in the rate of falls (31%).The secondary research questions will address other process outcomes to inform a larger trial and evaluate the effectiveness of the intervention on physical activity levels, physical performance, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Patients who do not exercise beyond moving around/walking during activities of daily living or exercise occasionally/during certain seasons more than others, and are interested in information about an exercise program offered by CFFM will be contacted about the study. To qualify for the study, patients must be: (i) 75 years or older, (ii) able to communicate in English (if unable to speak English, patient may qualify if a translator can attend program sessions and assist with completion of program materials), and (iii) able to give informed consent.

Exclusion Criteria:

Patients will be excluded if they: (i) currently participate in lower body muscle strengthening and balance exercise 3 or more times per week for 30 minutes or more, (ii) have a known diagnosis of dementia (those with mild cognitive impairment may be eligible if the can understand instructions or have a caregiver that can assist with the program) , (iii) have any significant lung disease, moderate to severe chronic obstructive pulmonary disease, and (iv) have contraindication(s) to exercise (e.g., uncontrolled hypertension).

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-06; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lora Giangregorio, PhD, Principal Investigator — University of Waterloo
Locations (1):
- Centre for Family Medicine, Kitchener, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lifestyle-integrated Functional Exercise
Started | 48
Enrolled in Intervention | 44
Completed | 32
Not Completed | 16
Not completed — Lost to Follow-up | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 13

BASELINE CHARACTERISTICS:
Population: Note: 1 participant did not agree to data collection for secondary outcomes.
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.6 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 18
Region of Enrollment [Number; unit: participants]
  Canada | 47

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment
Description: Feasibility of recruitment is defined as the number of participants recruited (feasibility) over six months.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 48
Participants | 48

2. Primary Outcome: Retention
Description: Retention is defined as the number of participants retained at Study Visit #1 (6-month follow-up).
Time Frame: 6 months
Population: Participants in the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 48
Participants | 32

3. Primary Outcome: Adherence (Including Withdrawals)
Description: Adherence is defined as the number of days each week that the participant completes/integrates strength and balance activities into daily tasks. Adherence will be 100% if participants complete the balance and strength activities at least 3 days per week.
Time Frame: 6 months
Population: Participants that enrolled in the intervention only
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 44
Participants
  Weeks 1-8 | 27
  Weeks 9-16 | 25
  Weeks 17-24 | 22

4. Secondary Outcome: Change in Physical Activity- Moderate-to-vigorous Physical Activity (MVPA) (Minutes/Week)
Description: * Participants will wear a physical activity monitor (Actigraph accelerometer) for seven days following Study Visit #1 (baseline) and Study Visit #2 (6 month follow-up) to determine the number of minutes spent sedentary and in light, moderate, and moderate-to-vigorous physical activity.
  * Participants will complete the IPAQ at Study Visit #1 (baseline) and Study Visit #2 (6 month follow-up) to evaluate changes in self-reported time spent performing physical activity.
Time Frame: Baseline, 6 months
Population: 21 participants completed accelerometer data collection at baseline and follow-up
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 32
minutes/week
  Accelerometer - MVPA - Baseline: number analyzed (Participants) | 21
  Accelerometer - MVPA - Baseline | 58.6 (111.1)
  Accelerometer - MVPA - 6 months: number analyzed (Participants) | 21
  Accelerometer - MVPA - 6 months | 52.5 (96.8)
  IPAQ - MVPA - Baseline | 41.2 (80.6)
  IPAQ - MVPA - 6 months | 60.6 (125.1)

5. Secondary Outcome: Change in Physical Performance- Scores on the Short Physical Performance Battery (SPPB)
Description: The SPPB consists of balance tests (side-by-side, semi-tandem, and tandem standing), gait speed during 4-meter walk test, and the average time taken to rise from a chair with arms folded across chest and sit back down (Five-Times-Sit-to-Stand test), sub-scores of which are added to determine a composite score (0-12), with higher scores indicative of better performance. Participants will complete physical performance tests as a measure of balance, mobility, and leg strength at Study Visits 1 (Baseline) and 2 (at 6 months).
Time Frame: Baseline, 6 months
Population: Note: 5 participants partially completed follow-up data collection (we administered questionnaire data over the phone because certain participants were unwilling to come to our centre for data collection) and therefore, SPPB data collection at baseline and 6-month follow-up was reported in 27 participants.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 27
score on a scale
  Baseline | 9.78 (1.97)
  6 months | 9.63 (2.26)

6. Secondary Outcome: Change in Quality of Life- EQ5D Dimensions and VAS Score
Description: Health-related quality of life will be assessed using the EQ5D health questionnaire at Study Visits 1 (Baseline) and 2 (at 6 months) to determine scores for all five dimensions (mobility, self-care, usual activities, pain/discomfort, and depression/anxiety) and the visual analogue scale (VAS). EQ5D VAS scores range 0-100, with higher scores indicating better overall health.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 32
units on a scale
  Baseline | 70.84 (14.15)
  6 months | 76.17 (14.44)

7. Secondary Outcome: Number of Falls
Description: Number of falls will be recorded daily on the postage-paid monthly diaries throughout the entire study (along with exercise information). A fall will be defined as an "a slip or a trip where the participant loses their balance and part or all of their body lands on the ground, floor or lower level".
Time Frame: 6 months
Population: Note: 1 participant did not agree to data collection for secondary outcomes
Measure: Number; unit: falls
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 47
falls | 19

8. Secondary Outcome: Number of Participants With Falls
Description: Number of participants with falls will be recorded daily on the postage-paid monthly diaries throughout the entire study (along with exercise information). A fall will be defined as an "a slip or a trip where the participant loses their balance and part or all of their body lands on the ground, floor or lower level".
Time Frame: 6 months
Population: Note: 1 participant did not agree to data collection for secondary outcomes
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 47
Participants | 10

9. Secondary Outcome: Number of Participants With Multiple Falls
Description: Number of participants with multiple falls will be recorded daily on the postage-paid monthly diaries throughout the entire study (along with exercise information). A fall will be defined as an "a slip or a trip where the participant loses their balance and part or all of their body lands on the ground, floor or lower level".
Time Frame: 6 months
Population: Note: 1 participant did not agree to data collection for secondary outcomes
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 47
Participants | 3

10. Secondary Outcome: Number of Participants With Adverse Events or Injuries (Serious or Otherwise)
Description: Participants will be instructed by the research coordinator and physiotherapist to report adverse events or injuries (serious or otherwise) to the research coordinator. Participants will be asked about illnesses or injuries at exercise sessions, follow-up phone calls, and Study Visit #2 (6 month follow-up). Intervention side effects (e.g., falls, fractures) and three types of adverse events will represent secondary outcomes (serious adverse events, adverse events possibly linked to the intervention, and adverse events that lead to study withdrawal or cessation of intervention).
Time Frame: 6 months
Population: Note: 1 participant did not agree to data collection for secondary outcomes
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 47
Participants
  Serious adverse events | 5
  Non-serious adverse events | 14

11. Secondary Outcome: Average Scores on Fidelity Rating Form - Individual and Group Sessions
Description: Fidelity evaluation of video-taped exercise sessions for first and last cohorts in the intervention (all sessions for first and last 4-5 individuals forming a group) will be conducted. A rating of physiotherapist compliance and participant uptake and descriptive feedback will be obtained. Fidelity rating forms (designed in-house by the study team) were filled out for the individual session (e.g., purpose and aims of LiFE program explained) and group sessions (e.g., PT demonstrated the activity to the group and identified situations to embed the activity). Each program criterion was scored out of 2 (0 = not done at all, 1 = done but could be better, 2 = done well) for 34 criteria for the individual session and for 17 criteria for the group sessions with any disagreement resolved via third-party.
Time Frame: 6 months
Population: Note: 1 participant did not agree to data collection for secondary outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 47
score on a scale
  Individual session | 1.8 (0.4)
  Group session | 1.9 (0.2)

12. Secondary Outcome: Sum of Scores on Fidelity Rating Forms - Individual and Group Sessions
Description: Fidelity evaluation of video-taped exercise sessions for first and last cohorts in the intervention (all sessions for first and last 4-5 individuals forming a group) will be conducted. A rating of physiotherapist compliance and participant uptake and descriptive feedback will be obtained. Fidelity rating forms (designed in-house by the study team) were filled out for the individual session (e.g., purpose and aims of LiFE program explained) and group sessions (e.g., PT demonstrated the activity to the group and identified situations to embed the activity). Each program criterion was scored out of 2 (0 = not done at all, 1 = done but could be better, 2 = done well) for 34 criteria for the individual session (sum of scores expressed out of 68) and 17 criteria for the group sessions (sum of scores expressed out of 34) with any disagreement resolved via third-party.
Time Frame: 6 months
Population: Note: 1 participant did not agree to data collection for secondary outcomes.
Measure: Number; unit: total score on a scale
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 47
total score on a scale
  Individual Session | 62
  Group Session | 33

13. Secondary Outcome: Number of Participants Who Provided Feedback on the Barriers and Facilitators to the Implementation of the Exercise Program
Description: Barriers and facilitators to implementation from the perspectives of the participants were identified using in-person or teleconference semi-structured interviews. Semi-structured interviews were conducted in-person with the participants at the 6-month follow-up time-point. The interviews with the participants included open-ended questions to understand their experience and level of satisfaction with the program (reasons for joining the program, observed benefits, areas for improvement, what they liked/disliked, general strategies for physical activity PA).
Time Frame: 6 months
Population: Note: 1 participant did not agree to data collection for secondary outcomes
Measure: Number; unit: participants
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 47
participants | 47

14. Secondary Outcome: Change in TFEQ-R21 Score- Cognitive Restraint Subscale
Description: The TFEQ-R21 questionnaire will be administered at Study Visit #1 (baseline), Exercise Session #1, and Study Visit #2 (6 month follow-up) as measures of eating behaviours, including cognitive restraint, uncontrolled eating, and emotional eating. The test-retest reliability of the TFEQ-R21 as a measure of eating behaviour in older adults aged 75 years or older will also be examined to determine consistency and stability of the instrument in the sample population. Subscale scores could range from 0 to 100 with higher scores indicating higher cognitive restraint.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 32
score on a scale
  Cognitive restraint score - Baseline | 16.0 (18.1)
  Cognitive restraint score - 6 months | 16.9 (20.9)

15. Secondary Outcome: Change in TFEQ-R21 Score - Uncontrolled Eating Subscale
Description: The TFEQ-R21 questionnaire will be administered at Study Visit #1 (baseline), Exercise Session #1, and Study Visit #2 (6 month follow-up) as measures of eating behaviours, including cognitive restraint, uncontrolled eating, and emotional eating. The test-retest reliability of the TFEQ-R21 as a measure of eating behaviour in older adults aged 75 years or older will also be examined to determine consistency and stability of the instrument in the sample population. Subscale scores could range from 0 to 100 with higher scores indicating higher uncontrolled eating behaviour.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 32
score on a scale
  Uncontrolled eating score - Baseline | 45.5 (30.0)
  Uncontrolled eating score - 6 months | 45.5 (23.5)

16. Secondary Outcome: Change in TFEQ-R21 Score - Emotional Eating Behaviour Subscale
Description: The TFEQ-R21 questionnaire will be administered at Study Visit #1 (baseline), Exercise Session #1, and Study Visit #2 (6 month follow-up) as measures of eating behaviours, including cognitive restraint, uncontrolled eating, and emotional eating. The test-retest reliability of the TFEQ-R21 as a measure of eating behaviour in older adults aged 75 years or older will also be examined to determine consistency and stability of the instrument in the sample population. Subscale scores could range from 0 to 100 with high scores indicating higher emotional eating behaviour.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 32
score on a scale
  Emotional eating score - Baseline | 15.5 (23.1)
  Emotional eating score - 6 months | 14.3 (20.6)

17. Other Pre Specified Outcome: Session Attendance
Description: Number of intervention sessions attended by participation
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 48
Participants
  Withdrew prior to program | 4
  1-2 sessions | 7
  3-4 sessions | 8
  5 sessions | 29

18. Post Hoc Outcome: Adherence (Excluding Withdrawals)
Description: as for outcome 3
Time Frame: 6 months
Population: Participants that enrolled in the intervention only
Measure: Count of Participants; unit: Participants
Arm/Group | Lifestyle-integrated Functional Exercise
Number analyzed (Participants) | 44
Participants
  Weeks 1-8 | 27
  Weeks 9-16: number analyzed (Participants) | 38
  Weeks 9-16 | 25
  Weeks 17-24: number analyzed (Participants) | 36
  Weeks 17-24 | 22

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Lifestyle-integrated Functional Exercise
Serious Adverse Events (participants affected / at risk) | 5/48
Other Adverse Events (participants affected / at risk) | 14/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle-integrated Functional Exercise (N=48)
Infection in big toe secondary to diabetes (Metabolism and nutrition disorders) | 1 (1) — Resulted in hospitalization
Worsening of COPD symptoms (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Resulted in hospitalization
Severe chest/abdominal pain (Cardiac disorders) | 1 (1) — Resulted in hospitalization
Diabetic episode (Metabolism and nutrition disorders) | 1 (1) — Resulted in hospitalization
Intracerebral hemorrhage (Vascular disorders) | 1 (1) — Resulted in death
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lifestyle-integrated Functional Exercise (N=48)
Heel pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to the intervention
Hamstring strain (Musculoskeletal and connective tissue disorders) | 1 (1) — Possibly related to the intervention
Pneumonia/flu (Infections and infestations) | 2 (2)
Chronic leg pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Fall-related injury (Injury, poisoning and procedural complications) | 2 (2)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Racing heart rate (Cardiac disorders) | 1 (1)
Strained rotator cuff (Musculoskeletal and connective tissue disorders) | 1 (1)
Hip tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Dementia diagnosis (Nervous system disorders) | 1 (1)
Heel spur (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes